CLINICAL TRIAL: NCT03278938
Title: Add-on to Cognitive, ERP and EEG Asymmetry in Affective Disorders (#6559R) [Formerly #5723]
Brief Title: Add-on to Cognitive, Event-Related Potentials (ERP) and Electroencephalogram (EEG) Asymmetry in Affective Disorders
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: PI Retired and no data was collected
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: #5723
Record Dates: First submitted 2013-05-16; First posted 2017-09-12 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Depressive Illness
Keywords: depression; citalopram; bupropion; combination therapy
MeSH Terms: conditions — Depression | interventions — Bupropion; Citalopram

STUDY DESIGN:
Intervention Model Description: treatment in this study was determined by treatment received in prior study; i.e., those who had received escitalopram then receive escitalopram + bupropion; those initially taking bupropion then receive escitalopram + bupropion
Oversight: Data Monitoring Committee: No

ARMS (2):
- bupropion added to citalopram (Active Comparator): patients who did not remit with citalopram will continue at the same dose and have bupropion added
  Interventions: Drug: bupropion; Drug: citalopram
- citalopram added to bupropion (Active Comparator): Patients who did not remit with bupropion will have bupropion continued at the same dose and citalopram will be added
  Interventions: Drug: bupropion; Drug: citalopram

INTERVENTIONS:
Drug: bupropion — FDA approved drug for treating depression
  Other Names: Wellbutrin
Drug: citalopram — FDA approved treatment for depression
  Other Names: Celexa

SUMMARY:
Depressed patients unremitted after monotherapy with citalopram or bupropion will remit following six weeks treatment with the combination of citalopram and bupropion.

DETAILED DESCRIPTION:
Participants in another study who did not remit during 12 weeks treatment with citalopram (to 40 mg/d) or bupropion (to 450 mg/d) will have citalopram (to 40 mg/d) or bupropion (to 450 mg/d) added for six weeks.

ELIGIBILITY:
Inclusion Criteria:

* non-remission in Protocol #6559R
* age 18-66
* signs informed consent
* physically healthy

Exclusion Criteria:

* bipolar disorder
* history of psychosis
* history of anorexia nervosa or bulimia
* history of seizure disorder, significant brain trauma or other medical reason to suspect increased seizure risk

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-06-29 (Estimated); Primary Completion 2016-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Hamilton Rating Scale | weeks 6
  Decrease in score for Hamilton Rating Scale for Depression, 17-item version

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan W Stewart, MD, Principal Investigator — Research Psychiatrist II at New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

REFERENCES:
- See also: web site for the Depression Evaluation Service, New York State Psychiatric Institute — http://www.depression-nyc.org